CLINICAL TRIAL: NCT01329861
Title: Guided Internet-based Cognitive Behavioural Treatment for Chronic Back Pain Reduces Catastrophizing:a Randomized Controlled Trial
Brief Title: Internet-based Cognitive Behavioural Treatment for Chronic Back Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Linkoeping University (Other Government)
Collaborators: Uppsala University (Other)
Responsible Party: Gerhard Andersson, professor, Linkoeping University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: smarta2011
Record Dates: First submitted 2011-04-04; First posted 2011-04-06 (Estimated); Last update posted 2011-04-06 (Estimated); Status verified 2011-04

CONDITIONS: Back Pain Lower Back Chronic
Keywords: chronic back pain; internet based treatment; pain management programme; cognitive behavioural therapy; minimal therapist contact

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Internet delivered CBT (Experimental): Internet delivered cognitive behavioral intervention, 8 weeks treatment.
  Interventions: Behavioral: Guided Internet-based cognitive behavioural treatment
- Control condition (No Intervention): Wait-list condition, received treatment after post-treatment assessment.

INTERVENTIONS:
Behavioral: Guided Internet-based cognitive behavioural treatment — Eight weeks internet-based cognitive behavioural treatment. Treatment consisted of education, cognitive skills acquisition, behavioural rehearsal, generalization and maintenance.
  Arms: Internet delivered CBT

SUMMARY:
The aim of this study was to investigate whether an Internet-based cognitive behavioural intervention would have an effect on the symptoms of chronic back pain.

DETAILED DESCRIPTION:
All participants were screened in a live, structured interview before inclusion. It´s a experimental design with a treatment and a control group measured before and after a treatment period.

ELIGIBILITY:
Inclusion Criteria:

* age between 18-65 years
* access to the Internet
* having been in contact with a physician
* back pain of chronic nature
* in current employment or on short-term sick leave(not longer than 6 months)

Exclusion Criteria:

* wheelchair user
* surgical treatment planned
* history of cardiovascular treatment
* severe depression

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2004-06; Primary Completion 2005-05 (Actual); Study Completion 2005-08 (Actual)

PRIMARY OUTCOMES:
Coping Strategies Questionnaire - catastrophizing subscale (CSQ) | Two weeks pre treatment to two weeks post treatment
  Change from baseline in the catastrophizing subscale to two weeks post treatment.

SECONDARY OUTCOMES:
Multidimensional Pain Inventory (MPI) | Change from baseline Two weeks pre treatment to two weeks post treatment
  MPI, assess psychosocial and behavioural consequences of pain. It´s divided into 2 sections and consisting of 8 scales. These are: Pain Severity, Interference, Life Control, Affective Distress, Support, Punishing Responses, Solicitous Responses and Distracting Responses.
Pain and Impairment Relationship Scale (PAIRS) | Change from baseline Two weeks pre treatment to two weeks post treatment.
  The questionnaire assesses beliefs and attitudes that patients have regarding pain and ability to function despite discomfort.
Hospital Anxiety and Depression Scale(HADS). | Change from baseline Two weeks pre treatment to two weeks post treatment.
  HADS is designed to measure anxiety and depression in non-psychiatric patients treated at hospital clinics.
Quality of Life Inventory (QOLI) | Change from baseline Two weeks pre treatment to two weeks post treatment.
  The assessment yields an overall score and profile for 16 areas of life: health, self-esteem, goals and values, money, work, play, learning, creativity, helping, love, friends, children, relatives, home, neighbourhood and community.

CONTACTS AND LOCATIONS:
Overall Officials: Gerhard Andersson, Professor, Study Director — Linkoeping University; Monica Buhrman, MSc, Principal Investigator — Uppsala University; Elisabeth Nilsson-Ihrfelt, MSc, Study Chair — Uppsala University; Maria Jannert, MSc, Study Chair — Linkoeping University; Lars Ström, PhD, Study Chair — Livanda (private practice) Västerås
Locations (1):
- Uppsala University, Uppsala, Sweden